CLINICAL TRIAL: NCT05944835
Title: Validation of Numerical Simulation to Predict Proximal Deployment of Standard Stents
Acronym: ProxSim
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0342
Record Dates: First submitted 2023-07-04; First posted 2023-07-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-07

CONDITIONS: Surgery
Keywords: Endoprosthesis; proximal neck; numerical simulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient who has been treated for an aortoiliac aneurysm: Any patient who has been treated for an aortoiliac aneurysm with a standard Medtronic Endurant aortic stent, standard Gore Excluder or conformable Gore Excluder
  Interventions: Other: Analyzed on the post-operative scanner

INTERVENTIONS:
Other: Analyzed on the post-operative scanner — Analyzed on the post-operative scanner

SUMMARY:
Endoprosthesis treatment of aortic pathologies has become the reference in the vast majority of situations. The success of this treatment is conditioned by the choice of the endoprosthesis which must be as adapted as possible to the anatomy. This choice is currently based on manual geometric measurements performed on the preoperative scanner using conventional image processing software.

The morphological result of the implantation of the endoprosthesis in the aorta is obtained by a CT scan carried out postoperatively. This scanner makes it possible to define the positioning of the endoprosthesis, the apposition surfaces between the aorta and the endoprosthesis and to predict the long-term result.

ELIGIBILITY:
Inclusion Criteria:

- Any patient who has been treated for an aortoiliac aneurysm with a standard Medtronic Endurant aortic stent, standard Gore Excluder or conformable Gore Excluder

Exclusion Criteria:

* Patient who has objected to the use of their data.
* No preoperative scanner available or insufficient injection quality
* Preoperative scanner with slice thickness greater than 3 mm

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient who has been treated for an aortoiliac aneurysm with a standard Medtronic Endurant aortic stent, standard Gore Excluder or conformable Gore Excluder
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
The accuracy of numerical simulation to predict the deployment at the level of the proximal neck of different types of standard stents used for the treatment of an aortoiliac aneurysm. | through study completion, an average of 1 year
  Wwill be evaluated by measuring the diameter and the position of the center of the first 3 simulated proximal stents will be compared to those of the real stents, analyzed on the post-operative scanner

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Louis Pradel, Bron, France